CLINICAL TRIAL: NCT07228624
Title: Expanding Use of Peri-Hematopoietic Cell Transplantation Ruxolitinib to Patients of Advanced Age With Myelofibrosis and Myelodysplastic Syndrome/Myeloproliferative Neoplasm Overlap Syndromes
Brief Title: Ruxolitinib Before, During and After Hematopoietic Cell Transplant in Older Patients With Myelofibrosis and Myelodysplastic Syndrome/Myeloproliferative Neoplasm Overlap Syndromes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125655; NCI-2025-07728 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020989 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic/Myeloproliferative Neoplasm; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Myelodysplastic-Myeloproliferative Diseases; Primary Myelofibrosis | interventions — ruxolitinib; Stem Cell Transplantation; Busulfan; Cyclophosphamide; fludarabine; Janus Kinase Inhibitors; Melphalan; Methotrexate; merphos; Tacrolimus; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib) (Experimental): PART 1: Patients receive ruxolitinib or alternate JAK-inhibitor for at least 8 weeks prior to the start of HCT conditioning.
  PART 2: Starting on day -4, patients receive ruxolitinib 5mg PO BID for 12 months then PO QD until 18 months. Patients receive high intensity conditioning with cyclophosphamide IV on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2 or reduced intensity conditioning with fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 15-30 minutes on days -3 and -2.
  Patients receive stem cells infusion on day 0. Starting on day -3, patients receive tacrolimus IV over 1-2 hours or PO every 12 hours for at least 100 days. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Additionally, patients undergo urine sample collection, echocardiography, and pulmonary function testing prior to conditioning and blood sample collection, bone marrow biopsy and aspiration, and spleen ultrasound or CT throughout the study.
  Interventions: Drug: Ruxolitinib; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Busulfan; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: JAK Inhibitor; Drug: Melphalan; Drug: Methotrexate; Drug: Tacrolimus; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy

INTERVENTIONS:
Drug: Ruxolitinib — Given PO
  Other Names: INCB 018424; INCB-018424; INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Given infusion
  Other Names: Allogeneic Hematopoietic Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: JAK Inhibitor — Given JAK inhibitor
  Other Names: JAK inhibitors; Janus Kinase Inhibitor
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow

SUMMARY:
This phase II trial tests the effect of adding ruxolitinib to standard graft versus host disease (GVHD) prevention in treating older patients with myelofibrosis (MF) or myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) overlap syndromes before, during, and after a donor (allogeneic) hematopoietic cell transplant (HCT). Allogeneic HCT is a procedure in which a person receives blood-forming stem cells (cells from which all blood cells develop) from a genetically similar, but not identical donor. Giving chemotherapy, such as cytoxan and busulfan or fludarabine and melphalan, before a donor transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. However, sometimes the transplanted cells from a donor can attack the body's normal cells (called GVHD). Giving standard prevention (prophylaxis) therapies, such as tacrolimus and methotrexate, after the transplant may stop this from happening. Methotrexate, a type of antifolate, is in a class of medications called antimetabolites. Methotrexate stops cells from using folic acid to make deoxyribonucleic acid and may kill cancer cells. Tacrolimus is used to help reduce the risk of rejection by the body of organ and bone marrow transplants. Ruxolitinib, a type of Janus-associated kinase (JAK) inhibitor, blocks a protein called JAK, which may help keep abnormal blood cells or cancer cells from growing. It may also lower the body's immune response and prevent the development of GVHD. Giving ruxolitinib before, during and after allogeneic HCT in addition to standard GVHD prophylaxis may be safe, tolerable and effective in preventing GVHD and improving outcomes in older patients with MF or MDS/MPN overlap syndrome.

DETAILED DESCRIPTION:
OUTLINE:

PART 1: Patients receive ruxolitinib or an alternate JAK-inhibitor for at least 8 weeks prior to the start of HCT conditioning. Starting on day -4, patients receive 5 mg of ruxolitinib orally (PO) twice daily (BID) for 12 months then PO once daily (QD) until 18 months. Patients receive high intensity conditioning with cyclophosphamide intravenously (IV) on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2 or reduced intensity conditioning with fludarabine IV over 30 minutes on days -6 to -2 and melphalan IV over 15-30 minutes on days -3 and -2.

PART 2: Patients receive stem cells infusion on day 0. Starting on day -3, patients receive tacrolimus IV over 1-2 hours or PO every 12 hours for at least 100 days. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Additionally, patients undergo urine sample collection, echocardiography, chest computed tomography (CT) and pulmonary function testing prior to conditioning and blood sample collection, bone marrow biopsy and aspiration and spleen ultrasound or CT at multiple time points before and after transplant.

After completion of study treatment, patients are followed at days 28, 100, 180, and at 9 months, 1 year, 18 months and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* PART 1 JAK INHIBITOR ADMINISTRATION: Age 18-75 years

  * Patients > 75 must be considered an HCT candidate, meet all protocol criteria and have comorbidity score =< 3 and Karnofsky performance status (KPS) > or = to 90. Patients. > 75 who do not meet these criteria may be presented at PCC for consensus exception
* PART 1 JAK INHIBITOR ADMINISTRATION: Disease criteria

  * Diagnosis of primary or secondary MF as defined by the 2022 World Health Organization classification system or the International Consensus Classification for Myeloid and Acute Leukemias
  * Diagnosis of an MDS/MPN overlap syndrome as defined by the 2022 World Health Organization
* PART 1 JAK INHIBITOR ADMINISTRATION: Ability to understand and the willingness to sign a written informed consent document
* PART 1 JAK INHIBITOR ADMINISTRATION: Patient must be a potential HCT candidate as assessed by the consenting physician
* PART 1 JAK INHIBITOR ADMINISTRATION: Patient must be agreeable to taking a JAK-inhibitor (ruxolitinib preferred) for at least 8 consecutive weeks immediately prior to conditioning and be willing to take ruxolitinib 5mg BID starting from day -4 prior to and continuing until 12 months post-transplant as tolerated followed by a 6-month taper.
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Meeting criteria for Part 1 at time of initiation of JAK-inhibitor, including the ability to understand and willingness to sign a written informed consent. Patients arriving to our institution for HCT and not enrolled in Part 1 may still be enrolled in Part 2 if Part 1 criteria are met. These patients will have Part 1 endpoints transcribed from their medical records
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Received a JAK-inhibitor for at least 8 weeks immediately prior to conditioning and be willing to take Rux from day -4 at the 5mg BID dose until 12 months post-transplant as tolerated followed by a 6 month taper
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Performance status score

  * Karnofsky ≥ 70 or > 90 for patients > 75 years old
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: HCT-CI Score < 8; if patient is > 75 years old HCT-CI < 3
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Calculated creatinine clearance using the Cockcroft-Gault formula or 24-hour urine creatinine clearance must be > 60 ml/min
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Total serum bilirubin must be < 3mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Transaminases must be < 3 x the upper limit of normal
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, and symptomatic biliary disease will be excluded
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Diffusion capacity of lung for carbon monoxide (DLCO) corrected > 60% normal. Patient may not be on oxygen
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Left ventricular ejection fraction > 40%
* DONOR: Human leukocyte antigen (HLA)-matched sibling donor
* DONOR: 10 of 10 HLA-matched unrelated donor
* DONOR: 9 of 10 allele or antigen mismatched unrelated donor
* DONOR: Peripheral blood is preferred over bone marrow
* DONOR: Matched unrelated donors may be preferred over siblings if the unrelated donor is < 30 years and the sibling is > 60 years. However, sibling donors < 70 should be preferred over mismatched unrelated donors

Exclusion Criteria:

* PART 1 JAK INHIBITOR ADMINISTRATION: Contraindication to receiving ruxolitinib including patients who have known hypersensitivity to JAK inhibitors and excipients
* PART 1 JAK INHIBITOR ADMINISTRATION: History of prior allogeneic transplant
* PART 1 JAK INHIBITOR ADMINISTRATION: Leukemic transformation (> 20% blasts)
* PART 1 JAK INHIBITOR ADMINISTRATION: Uncontrolled viral, bacterial, or fungal infection despite being on therapy
* PART 1 JAK INHIBITOR ADMINISTRATION: History of HIV infection
* PART 1 JAK INHIBITOR ADMINISTRATION: History of untreated tuberculosis (TB)
* PART 1 JAK INHIBITOR ADMINISTRATION: Pregnant or breastfeeding
* PART 1 JAK INHIBITOR ADMINISTRATION: Patients with history of myocardial infarction (MI), cerebrovascular accident (CVA) or unprovoked pulmonary embolism (PE)/deep vein thrombosis (DVT) in the past 6 months
* PART 1 JAK INHIBITOR ADMINISTRATION: Secondary malignancy in last 5 years with > 20% risk of relapse
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Contraindication to receiving ruxolitinib including patients who have known hypersensitivity to JAK inhibitors and excipients
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: History of prior allogeneic transplant
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Leukemic transformation (> 20% blasts)
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Uncontrolled viral or bacterial infection at the time of transplant data review and consent conference
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: History of HIV infection
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: History of untreated TB
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Requiring supplemental oxygen
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Pregnant or breastfeeding
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Secondary malignancy in last 5 years with > 20% risk of relapse
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Patients with a history of MI, CVA, or unprovoked PE/DVT in the past 6 months
* PART 2 ALLOGENEIC STEM CELL TRANSPLANT: Patients without an HLA-identical sibling donor, 10 of 10 HLA-matched or 9 of 10 mismatched unrelated donor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-21 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV graft versus host disease (GVHD) requiring systemic immune suppression | Up to day-100
  Will be estimated as a simple proportion, and the upper bound of the one-sided 95% confidence interval for the estimated proportion will be estimated using the Clopper-Pearson method. The exact binomial test will be used to compare the observed probability to the benchmark of 65%.

SECONDARY OUTCOMES:
Incidence of grade III-IV acute GVHD | Up to day-100
  Will be estimated as simple proportions and informally compared to the results from the historical cohort.
Incidence of any-grade chronic GVHD | Up to 1 and 2 years
  Will be treated as time-to-event endpoints, with specified point estimates.
Incidence of moderate-to-severe chronic GVHD | Up to 1 and 2 years
  Will be treated as time-to-event endpoints, with specified point estimates.
Non-relapse mortality (NRM) | At day-100
  Will be estimated as simple proportions and informally compared to the results from the historical cohort.
NRM | At 1 year
  Will be treated as time-to-event endpoints, with specified point estimates.
Remission status | At day-100
  Will be estimated as simple proportions and informally compared to the results from the historical cohort.
Relapse rate | At 1 and 2 years
  Will be treated as time-to-event endpoints, with specified point estimates.
Overall survival | Up to 1 year and by end of study, assessed up to 2 years
  Will be treated as time-to-event endpoints, with specified point estimates.
Incidence of graft failure | Up to day-100
  Will be estimated as simple proportions and informally compared to the results from the historical cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Salit, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No